CLINICAL TRIAL: NCT06966518
Title: Effectiveness of Intraoperative Combination of Ketamine and Magnesium Sulfate Infusions on Postoperative Analgesia in Patients Undergoing Open Rhinoplasty: A Randomized Controlled Trial
Brief Title: Intraoperative Combination of Ketamine and Magnesium Sulfate Infusions on Postoperative Analgesia in Open Rhinoplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sarah Ahmed, Lecturer of Anesthesia, Intensive care, and pain management, Faculty of Medicine, Ain Shams University, Cairo, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR1199/4/25
Record Dates: First submitted 2025-05-04; First posted 2025-05-12 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Intraoperative; Ketamine; Magnesium Sulfate; Postoperative Analgesia; Rhinoplasty
MeSH Terms: interventions — Ketamine; Magnesium Sulfate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KM Group (Experimental): Patients will receive a bolus of 0.5 mg/kg of ketamine given over a period of ten minutes followed by a constant infusion of 0.25 mg/kg/hr and a bolus dose of 30 mg/kg of magnesium sulfate during a 10-minute period followed by a continuous infusion of 9 mg/kg/hr.
  Interventions: Drug: Ketamine and Magnesium Sulfate
- Control group (Placebo Comparator): Patients will receive saline 0.9% as a control group.
  Interventions: Drug: Saline 0.9%

INTERVENTIONS:
Drug: Ketamine and Magnesium Sulfate — Patients will receive a bolus of 0.5 mg/kg of ketamine given over a period of ten minutes followed by a constant infusion of 0.25 mg/kg/hr and a bolus dose of 30 mg/kg of magnesium sulfate during a 10-minute period followed by a continuous infusion of 9 mg/kg/hr.
  Arms: KM Group
Drug: Saline 0.9% — Patients will receive saline 0.9% as a control group.
  Arms: Control group

SUMMARY:
The study aims to evaluate the effectiveness of intraoperative combination of ketamine and magnesium sulfate infusions on postoperative analgesia in patients undergoing open rhinoplasty.

DETAILED DESCRIPTION:
Postoperative pain remains one of the most crucial factors affecting patient satisfaction. These symptoms can be distressing for the patient and it may lead to negative psychological implications.

Ketamine is a non-competitive N-Methyl D-Aspartate (NMDA) receptor antagonist that works by blocking the NMDA receptors in the central and peripheral nervous systems.

Magnesium sulfate is also an antagonist for NMDA receptor that has been evaluated in several studies and showed that Mg sulfate decreased consumption of postoperative opioids.

Ketamine and magnesium sulfate have different sites of action on NMDA receptors, so their combination may produce a synergistic effect on NMDA receptors, resulting in more control of postoperative pain and more sparing of consumption of opioids.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years.
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status I - II.
* Scheduled for rhinoplasty under general anesthesia.

Exclusion Criteria:

* Receiving analgesic or any medications since 48 hours before the surgery.
* Drug addiction.
* Cardiovascular disease.
* Respiratory disease, renal, liver, metabolic and neurological disease.
* Pregnancy or breast feeding.
* Asthma.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Total morphine consumption | 24 hours postoperatively
  Rescue analgesia of morphine will be given as a 3 mg bolus if the numeric rating scale (NRS) > 3, to be repeated after 30 min if pain persists until the NRS < 4.

SECONDARY OUTCOMES:
Time to the 1st rescue analgesia. | 24 hours postoperatively
  Time to the first request for the rescue analgesia (time from end of surgery to first dose of morphine administrated).
Degree of pain | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the numeric rating scale (NRS). NRS (0 represents "no pain" while 10 represents "the worst pain imaginable"). NRS will be assessed at 0, 4, 6, 8, 12, 18, and 24 h postoperatively.
Heart rate | Till the end of surgery (Up to 2 hours)
  Heart rate will be recorded preoperatively and every 15 minutes till the end of surgery.
Mean arterial pressure | Till the end of surgery (Up to 2 hours)
  Mean arterial pressure will be recorded preoperatively and every 15 minutes till the end of surgery.
Degree of patient satisfaction | 24 hours postoperatively
  Degree of patient satisfaction will be assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied)
Incidence of adverse events. | 24 hours postoperatively
  Incidence of adverse events such as bradycardia, hypotension, nausea, vomiting, respiratory depression, hallucinations, nightmares, blurred vision, dizziness or any other complication.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.